CLINICAL TRIAL: NCT00050089
Title: CSP #512 - Options in Management With Anti-Retrovirals (OPTIMA), Management of Patients With HIV Infection for Whom First and Second-line Highly Active Anti-Retroviral Therapy Has Failed
Brief Title: CSP #512 - Options in Management With Anti-Retrovirals
Acronym: OPTIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Medical Research Council (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 512
Record Dates: First submitted 2002-11-20; First posted 2002-11-22 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: AIDS; HIV Infections
Keywords: AIDS; antiretrovirals; ART; drug-free period; HAART; HIV; human immunodeficiency virus; randomized; structured treatment interruptions
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No ARDFP+Standard-ART (Active Comparator): No Antiretroviral Drug-Free Period (No ARDFP) and Standard-ART
  Interventions: Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP; Drug: Standard ART vs Mega ART
- No ARDFP+Mega-ART (Active Comparator): No Antiretroviral Drug-Free Period (No ARDFP) and Mega-ART
  Interventions: Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP; Drug: Standard ART vs Mega ART
- ARDFP+Standard-ART (Active Comparator): Antiretroviral Drug-Free Period (ARDFP) and Standard-ART
  Interventions: Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP; Drug: Standard ART vs Mega ART
- ARDFP+Mega-ART (Active Comparator): Antiretroviral Drug-Free Period (ARDFP) and Mega-ART
  Interventions: Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP; Drug: Standard ART vs Mega ART

INTERVENTIONS:
Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP — Continuation or interruption of ART treatment
  Arms: No ARDFP+Standard-ART
Drug: Standard ART vs Mega ART — Standard therapy vs Intensified therapy
  Arms: No ARDFP+Standard-ART
Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP — Continuation or interruption of ART treatment
  Arms: No ARDFP+Mega-ART
Drug: Standard ART vs Mega ART — Standard therapy vs Intensified therapy
  Arms: No ARDFP+Mega-ART
Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP — Continuation or interruption of ART treatment
  Arms: ARDFP+Standard-ART
Drug: Standard ART vs Mega ART — Standard therapy vs Intensified therapy
  Arms: ARDFP+Standard-ART
Other: No Antiretroviral Drug-Free Period (No ARDFP) vs ARDFP — Continuation or interruption of ART treatment
  Arms: ARDFP+Mega-ART
Drug: Standard ART vs Mega ART — Standard therapy vs Intensified therapy
  Arms: ARDFP+Mega-ART

SUMMARY:
This 'pragmatic' trial is a 2X2 open randomized study of patients in advanced HIV disease who have failed on conventional Highly Active Antiretroviral Therapy (HAART) regimens including all three classes of anti-HIV drugs. The first randomization will allocate patients to an intended 3-month antiretroviral drug-free period (ARDFP) or No ARDFP. The second randomization will allocate patients to Mega-ART (5+ drugs) or to Standard-ART (up to 4 drugs). The total study duration is 6.5 years with 5 years of intake and 1.5 year (minimum) of follow-up; median duration of patient follow-up is about 4 years. The target sample size is 390 patients and will provide 75% power to detect a 30% reduction in the hazard rate for the primary endpoint with mega-ART. Sixty-four sites will be participating in the trial--24 VA, 19 UK and 21 Canada.

DETAILED DESCRIPTION:
Primary Hypothesis:

Compared to patients in Standard Antiretroviral Therapy (ART), patients in Mega-ART assuming full compliance, will experience a 30% reduction in the hazard of reaching a clinical endpoint (AIDS event or death).

Secondary Hypotheses:

Time to development of a new, non-HIV related serious adverse event, health related quality of life, the incidence of grade 3 or 4 clinical or laboratory adverse events and changes in virological and immunological markers (CD4 cell count, viral load, resistance profiles) will vary between the different treatment strategies.

Interventions:

Eligible patients will be randomized to one of four treatment strategy arms:

1. No Antiretroviral Drug-Free Period (No ARDFP) and Standard-ART
2. No Antiretroviral Drug-Free Period (No ARDFP) and Mega-ART
3. Antiretroviral Drug-Free Period (ARDFP) and Standard-ART
4. Antiretroviral Drug-Free Period (ARDFP) and Mega-ART

Note: The 'first' randomization will be ARDFP vs No ARDFP. Patients randomized to No ARDFP will receive their 'second' randomization at the same time. However, patients randomized to an Antiretroviral Drug Free Period (ARDFP) will receive their 'second' randomized assignment (Standard or Mega-ART) at the end of the ARDFP.

Note: All Serious Adverse Events were coded using the MedDRA coding dictionary; other (not serious) Adverse Events were collected as part of the study but were not coded using MedDRA or any other standardized coding dictionary.

This is the first trial of a Tri-National collaboration effort between the UK MRC, the Canadian CIHR and the VA CSP. The OPTIMA Trial was reviewed and approved by CSEC on October 12, 2000. The pre-kickoff meeting was held on March 21, 2001 in Washington, DC. The VA study kickoff meeting was held in Dallas, TX on May 16-18, 2001 and the Canadian kickoff was held in Toronto on May 29, 2001. The UK will have individual site initiation. As of October 17, 2005 there have been 357 patients enrolled in OPTIMA, at 64 sites in the three countries (279 in the VA, 41 in Canada and 37 in the UK). To date there are 64 sites actively participating in the study (24 in the VA, 19 in UK and 21 in Canada). Last date of patient follow-up was December 31, 2007.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Age of 18 years or more
* Serologic or virologic diagnosis of HIV infection
* Failure of at least two different multi-drug regimens that include drugs of all 3 classes that the patient can tolerate or laboratory evidence of resistance to drugs in each of the 3 classes
* Had at least 3 months of current ART and are still on treatment
* Two most recent results (which can include screening) on current ART of CD4 count less than or equal to 300 cells/mm3 or less than or equal to 15%, and a plasma viral load greater than or equal to 5,000 copies/ml (Roche Amplicor, v1.0), or greater than or equal to 2,500 copies/ml (by bDNA: Bayer v3.0/Chiron v3.0 or PCR:Roche Amplicor Monitor/COBAS v1.5)

Exclusion Criteria:

* Pregnancy, breast-feeding or planned pregnancy
* Likelihood of poor protocol follow-up or if Mega-Art is not feasible (due to significant intolerance of many ARV drugs)
* Serious, uncontrolled major opportunistic infection (OI) within 14 days of screening
* Likelihood of early death due to non-HIV disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2001-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Brown, Study Chair — VA Medical Center, Bronx
Locations (30):
- United States (29):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Medical Center, Miami, Miami, Florida
  - Bay Pines VAMC (111J), St. Petersburg, Florida
  - West Palm Beach VA Medical Center, West Palm Beach, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Bronx, The Bronx, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - WJB Dorn Veterans Hospital, Columbia, Columbia, South Carolina
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
- VA Medical Center, San Juan, San Juan, Puerto Rico

REFERENCES:
- [Background] Kyriakides TC, Babiker A, Singer J, Cameron W, Schechter MT, Holodniy M, Brown ST, Youle M, Gazzard B; OPTIMA Study Team. An open-label randomized clinical trial of novel therapeutic strategies for HIV-infected patients in whom antiretroviral therapy has failed: rationale and design of the OPTIMA Trial. Control Clin Trials. 2003 Aug;24(4):481-500. doi: 10.1016/s0197-2456(03)00029-1. PMID 12865041
- [Background] Bedimo R, Kyriakides T, Brown S, Weidler J, Lie Y, Coakley E, Holodniy M. Predictive value of HIV-1 replication capacity and phenotypic susceptibility scores in antiretroviral treatment-experienced patients. HIV Med. 2012 Jul;13(6):345-51. doi: 10.1111/j.1468-1293.2011.00981.x. Epub 2012 Jan 26. PMID 22276745
- [Background] Kyriakides TC, Babiker A, Singer J, Piaseczny M, Russo J. Study conduct, monitoring and data management in a trinational trial: the OPTIMA model. Clin Trials. 2004;1(3):277-81. doi: 10.1191/1740774504cn022oa. PMID 16279253
- [Background] Dau B, Ayers D, Singer J, Harrigan PR, Brown S, Kyriakides T, Cameron DW, Angus B, Holodniy M. Connection domain mutations in treatment-experienced patients in the OPTIMA trial. J Acquir Immune Defic Syndr. 2010 Jun;54(2):160-6. doi: 10.1097/QAI.0b013e3181cbd235. PMID 20130473
- [Background] Bansback N, Sun H, Guh DP, Li X, Nosyk B, Griffin S, Barnett PG, Anis AH; OPTIMA TEAM. Impact of the recall period on measuring health utilities for acute events. Health Econ. 2008 Dec;17(12):1413-9. doi: 10.1002/hec.1351. PMID 18404664
- [Background] Desai S, Kyriakides T, Holodniy M, Al-Salman J, Griffith B, Kozal M. Evolution of genotypic resistance algorithms and their impact on the interpretation of clinical trials: an OPTIMA trial substudy. HIV Clin Trials. 2007 Sep-Oct;8(5):293-302. doi: 10.1310/hct0805-293. PMID 17956830
- [Result] Barnett PG, Chow A, Joyce VR, Bayoumi AM, Griffin SC, Nosyk B, Holodniy M, Brown ST, Sculpher M, Anis AH, Owens DK. Determinants of the cost of health services used by veterans with HIV. Med Care. 2011 Sep;49(9):848-56. doi: 10.1097/MLR.0b013e31821b34c0. PMID 21610542
- [Result] Nosyk B, Sun H, Bansback N, Guh DP, Li X, Barnett P, Bayoumi A, Griffin S, Joyce V, Holodniy M, Owens DK, Anis AH. The concurrent validity and responsiveness of the health utilities index (HUI 3) among patients with advanced HIV/AIDS. Qual Life Res. 2009 Sep;18(7):815-24. doi: 10.1007/s11136-009-9504-0. Epub 2009 Jun 27. PMID 19562514
- [Result] Anis AH, Nosyk B, Sun H, Guh DP, Bansback N, Li X, Barnett PG, Joyce V, Swanson KM, Kyriakides TC, Holodniy M, Cameron DW, Brown ST; OPTIMA Team1. Quality of life of patients with advanced HIV/AIDS: measuring the impact of both AIDS-defining events and non-AIDS serious adverse events. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):631-9. doi: 10.1097/QAI.0b013e3181a4f00d. PMID 19430303
- [Result] Joyce VR, Barnett PG, Bayoumi AM, Griffin SC, Kyriakides TC, Yu W, Sundaram V, Holodniy M, Brown ST, Cameron W, Youle M, Sculpher M, Anis AH, Owens DK. Health-related quality of life in a randomized trial of antiretroviral therapy for advanced HIV disease. J Acquir Immune Defic Syndr. 2009 Jan 1;50(1):27-36. doi: 10.1097/QAI.0b013e31818ce6f3. PMID 19295332
- [Result] Joyce VR, Barnett PG, Chow A, Bayoumi AM, Griffin SC, Sun H, Holodniy M, Brown ST, Kyriakides TC, Cameron DW, Youle M, Sculpher M, Anis AH, Owens DK. Effect of treatment interruption and intensification of antiretroviral therapy on health-related quality of life in patients with advanced HIV: a randomized, controlled trial. Med Decis Making. 2012 Jan-Feb;32(1):70-82. doi: 10.1177/0272989X10397615. Epub 2011 Mar 7. PMID 21383086
- [Derived] Holodniy M, Brown ST, Cameron DW, Kyriakides TC, Angus B, Babiker A, Singer J, Owens DK, Anis A, Goodall R, Hudson F, Piaseczny M, Russo J, Schechter M, Deyton L, Darbyshire J; OPTIMA Team. Results of antiretroviral treatment interruption and intensification in advanced multi-drug resistant HIV infection from the OPTIMA trial. PLoS One. 2011 Mar 31;6(3):e14764. doi: 10.1371/journal.pone.0014764. PMID 21483491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 368 participants were enrolled in the trial: 41 in Canada, 39 in the UK and 288 in the US-VA.
Pre-assignment Details: 339 participants were randomized to factorial design(Canada=41;UK=10;US-VA=288). 29 participants in the UK were enrolled in a protocol-approved option, where they were allowed to select one of the factors and be randomized to the other. All 29 selected the ARDFP vs No ARDFP factor and were randomized to the Standard-ART vs Mega-ART factor.
Groups:
- No ARDFP+Standard-ART: No Antiretroviral Drug-Free Period (No ARDFP) and Standard-ART
  Standard-ART: up to 4 anti-HIV drugs
- No ARDFP+Mega-ART: No Antiretroviral Drug-Free Period (No ARDFP) and Mega-ART
  Mega-ART: 5 or more anti-HIV drugs
- ARDFP+Standard-ART: Antiretroviral Drug-Free Period (ARDFP) and Standard-ART
  Intended duration of ARDFP: 12 week2 Standard-ART: up to 4 anti-HIV drugs
- ARDFP+Mega-ART: Antiretroviral Drug-Free Period (ARDFP) and Mega-ART
  Intended duration of ARDFP: 12 weeks Mega-ART: 5 or more anti-HIV drugs
Period: Overall Study
Arm/Group | No ARDFP+Standard-ART | No ARDFP+Mega-ART | ARDFP+Standard-ART | ARDFP+Mega-ART
Started | 106 | 98 | 86 | 78
Baseline | 91 (15 participants randomized in the UK Option scheme (not displayed in the 2X2 baseline data)) | 84 (14 participants randomized in the UK Option scheme (not shown in 2X2 baseline data)) | 86 | 78
Completed | 106 (For primary outcome assessment) | 98 (For primary outcome assessment) | 86 (For primary outcome assessment) | 78 (For primary outcome assessment)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: HIV-positive patients with a CD4 count <=300 cells/ul who had prior anti-retroviral treatment failure requiring retreatment
Groups:
- No ARDFP + Standard ART: Standard Antiretroviral Treatment regimen
- No ARDFP + Mega ART: Intensive Antiretroviral Treatment regimen
- ARDFP + Standard ART: Antiretroviral Treatment Interruption and Standard ART
- ARDFP + Mega ART: Antiretroviral Treatment Interruption and Intensive ART
- Total: Total of all reporting groups
Arm/Group | No ARDFP + Standard ART | No ARDFP + Mega ART | ARDFP + Standard ART | ARDFP + Mega ART | Total
Number analyzed (Participants) | 91 | 84 | 86 | 78 | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (8.99) | 48.3 (7.92) | 49.2 (8.1) | 48.2 (8.58) | 48.6 (8.39)
Age, Customized [Number; unit: participants]
  31-40 years | 16 | 11 | 12 | 15 | 54
  41-50 years | 35 | 41 | 36 | 30 | 142
  51-60 years | 33 | 28 | 31 | 28 | 120
  >60 years | 7 | 4 | 7 | 5 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 7
  Male | 90 | 82 | 84 | 76 | 332
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 45 | 38 | 35 | 160
  Black | 41 | 30 | 36 | 31 | 138
  Asian | 1 | 0 | 0 | 0 | 1
  Hispanic | 6 | 9 | 9 | 12 | 36
  Aboriginal | 1 | 0 | 1 | 0 | 2
  Other | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 77 | 71 | 73 | 67 | 288
  United Kingdom | 2 | 2 | 3 | 3 | 10
  Canada | 12 | 11 | 10 | 8 | 41
log10 Viral Load [Mean (Standard Deviation); unit: log10 copies/mL] | 4.76 (0.55) | 4.75 (0.76) | 4.64 (0.67) | 4.7 (0.75) | 4.71 (0.68)
CD4 cells/mm3 [Mean (Standard Deviation); unit: cells/mm^3] | 136 (112) | 127 (107) | 130 (106) | 127 (106) | 130 (108)
CD4 level [Number; unit: participants]
  CD4 <=100 cells/mm^3 | 38 | 38 | 36 | 33 | 145
  CD4 >100 cells/mm^3 | 53 | 46 | 50 | 45 | 194
Mode of HIV Infection [Number; unit: participants]
  Blood | 12 | 7 | 8 | 7 | 34
  Heterosexual | 20 | 19 | 22 | 19 | 80
  Intravenous Drug Use (IVDU) | 11 | 16 | 15 | 9 | 51
  Men who have Sex with Men (MSM) | 42 | 37 | 37 | 39 | 155
  Other | 6 | 5 | 2 | 4 | 17
  Unknown | 0 | 0 | 2 | 0 | 2
AIDS at entry [Number; unit: participants] — History of AIDS event at study entry
  participants
    Yes | 59 | 46 | 44 | 51 | 200
    No | 32 | 38 | 42 | 27 | 139
Hepatitis B (HBsAg) [Number; unit: participants]
  Yes | 10 | 4 | 15 | 8 | 37
  No | 81 | 80 | 71 | 70 | 302
Hepatitis C (Hep C anti-HCV) [Number; unit: participants]
  Yes | 17 | 21 | 27 | 12 | 77
  No | 74 | 63 | 59 | 66 | 262
OI medications for prophylaxis [Number; unit: participants] — Opportunistic Infections medications for prophylaxis at study entry
  participants
    Anti-PCP | 75 | 67 | 71 | 62 | 275
    Anti-CMV | 2 | 0 | 2 | 0 | 4
    Antibacterial | 43 | 39 | 33 | 37 | 152
    Antifungal | 22 | 23 | 22 | 19 | 86
Concomitant Medications [Number; unit: participants] — Not all study participants were on other Concomitant Medications. Numbers provided represent participants on those medications at baseline.
  participants
    Lipid Lowering | 24 | 20 | 33 | 21 | 98
    Other antiviral | 43 | 30 | 30 | 33 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New or Recurrent AIDS Event, or Death
Description: New or recurrent AIDS event or Death were compared between Standard-ART (standard) and Mega-ART (intensification)
Time Frame: From date of randomization until onset of primary outcome or end of study follow-up (12/31/2007) whichever occured first, up to 6.5 years
Population: This includes participants randomized to Standard-ART or Mega-ART (339 via the 2X2 factorial design and 29 via the UK Option Scheme)
Measure: Number; unit: participants
Groups:
- Standard-ART: This includes participants randomized to Standard-ART (No ARDFP+Standard-ART or ARDFP+Standard-ART)
- Mega-ART: This includes participants randomized to Mega-ART (No ARDFP+Mega-ART or ARDFP+Mega-ART)
Arm/Group | Standard-ART | Mega-ART
Number analyzed (Participants) | 192 | 176
participants | 83 | 82
Statistical Analysis 1: Comparison: Standard-ART vs Mega-ART; Time-to-event (Kaplan-Meier) and stratified log-rank test was used for the comparison; Test type: Superiority or Other; p = 0.69, Log Rank; Hazard Ratio (HR) = 1.165, 95% CI 2-sided [0.856 to 1.585] — The comparison was Mega-ART (intensification) vs Standard-ART (standard)

2. Primary Outcome: Number of Participants With New or Recurrent AIDS Event, or Death
Description: New or recurrent AIDS event or Death were compared between No ARDFP (continuation) and ARDFP (interruption)
Time Frame: as for outcome 1
Population: This includes participants randomized to No ARDFP or ARDFP (339 via the 2X2 factorial design and 0 via the UK Option Scheme)
Measure: Number; unit: participants
Groups:
- ARDFP: This includes participants randomized to ARDFP (ARDFP+Standard-ART or ARDFP+Mega-ART)
- No ARDFP: This includes participants randomized to No ARDFP (No ARDFP+Standard-ART or No ARDFP+Mega-ART)
Arm/Group | ARDFP | No ARDFP
Number analyzed (Participants) | 164 | 175
participants | 70 | 87
Statistical Analysis 1: Comparison: ARDFP vs No ARDFP; Time-to-event (Kaplan-Meier) and stratified log-rank analysis was performed; Test type: Superiority or Other; p = 0.49, Log Rank; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.674 to 1.275] — The comparison was ARDFP (interruption) vs No ARDFP (continuation)

3. Primary Outcome: Number of Participants With New or Recurrent AIDS Event, or Death
Description: New or recurrent AIDS event or Death were compared between No ARDFP (continuation)+Standard-ART (standard), No ARDFP (continuation)+Mega-ART (intensification), ARDFP (interruption)+Standard-ART (standard) and ARDFP (interruption)+Mega-ART (intensification)
Time Frame: as for outcome 1
Population: This includes participants randomized to one of the four interventions (339 via the 2X2 factorial design)
Measure: Number; unit: participants
Groups:
- No ARDFP + Standard ART: Standard ART regimen, with no prior ART interruption
- No ARDFP + Mega ART: Intensive ART regimen, with no prior ART interruption
- ARDFP + Standard ART: Standard ART regimen following ART interruption
- ARDFP + Mega ART: Intensive ART following ART interruption
Arm/Group | No ARDFP + Standard ART | No ARDFP + Mega ART | ARDFP + Standard ART | ARDFP + Mega ART
Number analyzed (Participants) | 91 | 84 | 86 | 78
participants | 46 | 41 | 35 | 35
Statistical Analysis 1: Comparison: No ARDFP + Standard ART vs No ARDFP + Mega ART vs ARDFP + Standard ART vs ARDFP + Mega ART; Stratified Log-rank test was used to compare the four treatment; Test type: Superiority or Other; p = 0.87, Log Rank

4. Secondary Outcome: Number of Participants With a New, Non-HIV Related Serious Adverse Event
Description: New, on-study non-HIV related Serious Adverse events were compared between Standard-ART (standard) and Mega-ART (intensification)
Time Frame: From date of randomization until onset of secondary outcome or end of study follow-up (12/31/2007) whichever occured first, up to 6.5 years
Measure: Number; unit: participants
Arm/Group | Standard-ART | Mega-ART
Number analyzed (Participants) | 192 | 176
participants | 97 | 88
Statistical Analysis 1: Comparison: Standard-ART vs Mega-ART; Time-to-event (Kaplan-Meier) and stratified log-rank test was used for the comparison; Test type: Superiority or Other; p = 0.92, Log Rank; Hazard Ratio (HR) = 1.008, 95% CI 2-sided [0.75 to 1.35] — The comparison was Standard-ART (standard) vs Mega-ART (intensification)

5. Secondary Outcome: Number of Participants With New, Non-HIV Related Serious Adverse Event
Description: New, on-study non-HIV related Serious Adverse events were compared between ARDFP (interruption) and No ARDFP (continuation)
Time Frame: as for outcome 4
Measure: Number; unit: participants
Arm/Group | ARDFP | No ARDFP
Number analyzed (Participants) | 164 | 175
participants | 84 | 92
Statistical Analysis 1: Comparison: ARDFP vs No ARDFP; Time-to-event (Kaplan-Meier) and stratified log-rank test was used for the comparison; Test type: Superiority or Other; p = 0.68, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.8 to 1.46] — The comparison was ARDFP (interruption) vs No ARDFP (continuation) of ART

ADVERSE EVENTS:
Description: MedDRA was used to code SAE of participants randomized to the 2x2 factorial design (n=339).Hence the number at risk for the four arms reflects only participants enrolled in the 2x2 factorial. Not Serious Adverse events were not coded using MedDRA.
Arm/Group | No ARDFP + Standard ART | No ARDFP + Mega ART | ARDFP + Standard ART | ARDFP + Mega ART
Serious Adverse Events (participants affected / at risk) | 55/91 | 56/84 | 54/86 | 49/78
Other Adverse Events (participants affected / at risk) | 0/106 | 0/98 | 0/86 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No ARDFP + Standard ART (N=91) | No ARDFP + Mega ART (N=84) | ARDFP + Standard ART (N=86) | ARDFP + Mega ART (N=78)
Acquired methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anaemia NOS (Blood and lymphatic system disorders) | 5 (7) | 5 (6) | 6 (10) | 5 (6)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Bone marrow depression NOS (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Secondary anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 1 (2) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia NOS (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder NOS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure NOS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (3) | 3 (3) | 0 (0) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiomyopathy NOS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiovascular disorder NOS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery atherosclerosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease NOS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Endocarditis NOS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia NOS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency NOS (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Retinitis NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis NOS (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vision abnormal NOS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain NOS (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Caecitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea NOS (Gastrointestinal disorders) | 5 (5) | 4 (5) | 4 (4) | 1 (1)
Diverticulitis NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal disorder NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Oesophagitis NOS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis NOS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Perirectal abscess (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting NOS (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0) | 2 (3)
Adverse drug reaction NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chest pain (General disorders) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Death NOS (General disorders) | 5 (5) | 0 (0) | 7 (7) | 6 (6)
Drug interaction NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation NOS (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrosis NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 7 (7) | 1 (4) | 3 (3) | 3 (4)
Weakness (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis NOS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic disorder NOS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis NOS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice NOS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity NOS (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immune reconstitution syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess NOS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acquired immunodeficiency syndrome NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arterio-venous fistula infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspergillosis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis bacterial NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 4 (4) | 2 (2)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central nervous system infection NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection NOS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Colitis pseudomembranous (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cryptococcosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus retinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epidural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
External ear infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection syphilitic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral NOS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gram-positive bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIV wasting syndrome (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 4 (4)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes viral infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Herpetic stomatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Histoplasmosis disseminated (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infected insect bite (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection NOS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis bacterial NOS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Meningitis viral NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Methicillin-resistant staphylococcal aureus infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (4)
Mucormycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium avium complex (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (3)
Necrotising fasciitis NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 2 (3) | 3 (7) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis NOS (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Otitis media acute NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parvovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Penile abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perianal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis carinii pneumonia (Infections and infestations) | 6 (8) | 7 (8) | 6 (7) | 5 (8)
Pneumonia NOS (Infections and infestations) | 6 (9) | 9 (12) | 9 (11) | 4 (4)
Pneumonia bacterial NOS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Pseudomonas aeruginosa infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyomyositis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection NOS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Scrotal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis MRSA (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Sepsis NOS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Septicaemia gram-positive (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Septicaemia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septicaemia salmonella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue abscess NOS (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Skin fungal infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toxoplasmosis NOS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection viral NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection NOS (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rash NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose NOS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Shunt malfunction NOS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound NOS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acid fast stain positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biopsy NOS (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laboratory test abnormal NOS (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function tests NOS abnormal (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (4) | 0 (0) | 1 (1)
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis NOS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal canal cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic neoplasm malignant NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's disease NOS stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 1 (3) | 1 (1)
Laryngeal cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rectal cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
T-cell lymphoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsions NOS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dementia NOS (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine NOS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neurological findings abnormal NOS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral neuropathy aggravated (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subacute combined cord degeneration (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0) | 2 (2)
Tonic clonic movements (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug addiction (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Mood disorder NOS (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polysubstance dependence (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Psychotic disorder NOS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pre-renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus renal NOS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic cystitis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure NOS (Renal and urinary disorders) | 3 (3) | 2 (3) | 2 (2) | 3 (4)
Renal failure acute (Renal and urinary disorders) | 3 (6) | 2 (2) | 0 (0) | 3 (3)
Renal failure acute on chronic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment NOS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Testicular torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hilar lymphadenopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Pulmonary hypertension NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucocutaneous ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug abuser NOS (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Treatment noncompliance (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterio-venous fistula operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood product transfusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemodialysis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal fistula repair (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Stent insertion NOS (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction NOS (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Arterio-venous fistula thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atherosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep venous thrombosis NOS (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Haemorrhage NOS (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension aggravated (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension NOS (Vascular disorders) | 4 (5) | 0 (0) | 0 (0) | 3 (3)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis deep limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No